CLINICAL TRIAL: NCT06104566
Title: A Global Multicenter, Open Label, Randomized Phase 3 Registrational Study of Lisaftoclax (APG-2575) in Previously Treated Patients With Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (GLORA Study)
Brief Title: Global Trial in APG2575 for Patients With CLL/SLL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG2575CG301
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: CLL/SLL

STUDY DESIGN:
Intervention Model Description: 1:1 ratio to investigational arm (lisaftoclax in combination with BTKi ) or the control arm (BTKi).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Combination therapy
  Interventions: Drug: lisaftoclax +BTK inhibitor
- Arm 2 (Active Comparator): mono therapy
  Interventions: Drug: BTK inhibitor

INTERVENTIONS:
Drug: lisaftoclax +BTK inhibitor — lisaftolax + BTK inhibitor
  Arms: Arm 1
Drug: BTK inhibitor — BTK inhibitor
  Arms: Arm 2

SUMMARY:
This is a global multicenter, open label, randomized, registrational phase III study to investigate the efficacy and safety of lisaftoclax in combination with BTK inhibitors in CLL/SLL patients who previously treated with BTK inhibitors

DETAILED DESCRIPTION:
Approximately 440 patients will be enrolled, the patients who meet the eligibility criteria will be randomized in a 1:1 ratio to investigational arm (lisaftoclax in combination with a BTK inhibitor) or the control arm (BTK inhibitor alone). These patients with CLL/SLL have been on BTKi monotherapy and meet all other protocol required eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

1. - Age ≥ 18 years.
2. . Patients that have documented CLL/SLL who meet iwCLL 2018 criteria for CLL treatment guidelines are eligible for treatment and must be receiving BTKi monotherapy for at least 12 months
3. ECOG Performance Status grade 0-2
4. Adequate bone marrow function independent of growth factor or transfusion support within 2 weeks of screening initiation as follows:

   * Absolute neutrophil count ≥ 1.0 × 109/L
   * Platelet counts ≥ 75 × 109/L; in cases of thrombocytopenia
   * Total hemoglobin ≥ 9 g/dL,
5. Adequate renal function

   * Creatinine clearance must be > 50 ml/min directly measured with 24hr urine collection or calculated according to the modified formula of Cockcroft and Gault (for men: GFR ≈ ((140 - age) x actual body weight)/(72 x creatinine), for women x 0.85) or an equally accurate method.
   * For patients with creatinine values within the normal range, the calculation of clearance is not necessary. Dehydrated patients with an estimated creatinine clearance less than 50 ml/min may be eligible if a repeat estimate after adequate hydration is > 50 ml/min.
6. Adequate liver function as indicated by:

   * Total bilirubin ≤ 1.5 x ULN, except patients with known Gilbert's Syndrome
   * Aspartate aminotransferase (AST) ≤ 2.5 x the institutional ULN value
   * Alanine aminotransferase (ALT) ≤ 2.5 x the institutional ULN value,
   * International normalized Ratio (INR), Prothrombin Time (PT) or Activated Partial Thromboplastin time (APTT) ≤ 1.5×ULN.
7. Ability and willingness to provide written informed consent and to adhere to the study visit schedule and other protocol requirements

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 12 months
  To evaluate the progression-free survival (PFS) of lisaftoclax in combination with BTKi compared with BTKi monotherapy in CLL/SLL patients previously treated with BTKi as determined by independent radiological review committee (IRC) using the iwCLL guidelines

SECONDARY OUTCOMES:
overall survival | 12 months
  To evaluate overall survival (OS) of lisaftoclax in combination with BTKi versus BTKi

CONTACTS AND LOCATIONS:
Locations (2):
- MD Anderson Cancer Center, Houston, Texas, United States
- Kaluga Regional Clinical Research, Kaluga, Russia